CLINICAL TRIAL: NCT04623424
Title: Intestinal Microbiota Alteration by Antibiotics Used During Stem Cell Transplant Admission
Brief Title: Intestinal Microbiota in Stem Cell Transplant Transplant Admission
Status: Recruiting | Type: Observational
Sponsor: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, Shatha Farhan, Clinical Assistant Professor, Henry Ford Health System
Other Study IDs: 14270
Record Dates: First submitted 2020-11-03; First posted 2020-11-10 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Stem Cell Transplant Complications
MeSH Terms: interventions — Gastrointestinal Microbiome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: intestinal microbiota — Stoll samples will be tested for different bacteria

SUMMARY:
In this prospective study, the primary objective will be to investigate the association between the use of antibiotics administered during the admission period of Stem cell transplant (SCT) and the rate of overall change in microbiota composition across adjacent samples in time.

DETAILED DESCRIPTION:
Early preclinical studies suggested that intestinal microflora contribute to aGVHD and may be relapse. There is increasing evidence that use of antibiotics may have a detrimental impact on intestinal microbiota composition and, consequently, the outcome of SCT.However, effect on different antibiotic prophylaxis regimens and broad-spectrum antibiotics used during transplant and the intestinal microbiota composition and hence adverse outcomes are not known. Stool samples will be collected from patients who are undergoing SCT at:

1. preconditioning
2. at day 0 (stem cell infusion)
3. once in the period of day + 7-10 post SCT
4. once first day or second day of BMT OPD clinic visit
5. once if they develop >=grade I GVHD
6. once at time of recovery from GVHD

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-80 years
* patients undergoing allogenic or autologous SCT for malignant hematological conditions or bone marrow failure

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: stem cell transplant patients
Sampling Method: Non-Probability Sample
Enrollment: 255 (Estimated)
Dates: Start 2020-11-03 (Actual); Primary Completion 2026-11-03 (Estimated); Study Completion 2026-11-03 (Estimated)

PRIMARY OUTCOMES:
Changes in microbiome | Up to 6 months post stem cell transplant

CONTACTS AND LOCATIONS:
Overall Officials: shatha farhan, Principal Investigator — Henry Ford
Locations (1):
- Henry Ford Health System, Detroit, Michigan, United States